CLINICAL TRIAL: NCT04049253
Title: The Causal Connection Between Sng and Muscle Acidosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, Jiann-Her,Lin, Attending physician, Taipei Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: N201902030
Record Dates: First submitted 2019-07-23; First posted 2019-08-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Muscle Acidosis
Keywords: sngceptin; soreness; muscle acidosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acidic phosphate buffer solution (Experimental): pH5.2 phosphate buffer solution
  Interventions: Drug: Phosphate Buffer Solution
- Neutral phosphate buffer solution (Placebo Comparator): pH7.4 phosphate buffer solution
  Interventions: Drug: Phosphate Buffer Solution

INTERVENTIONS:
Drug: Phosphate Buffer Solution — Phosphate-buffered saline (abbreviated PBS) is a buffer solution commonly used in biological research. It is a water-based salt solution containing disodium hydrogen phosphate, sodium dihydrogen phosphate. The buffer helps to maintain a constant pH. The osmolarity and ion concentrations of the solutions match those of the human body (isotonic).
  Other Names: Sodium phosphate solution; Phosphate buffered saline

SUMMARY:
This proposed study suggests that peripheral tissue acidosis sensed by the somatosensory system (sngceptin) would evoke the sng perception in the brain. This hypothesis is based on investigators preliminary data that the peripheral muscle acidosis will evoked the central sng perception. This proposed study also identify the detection of brain activation areas related to the peripheral muscle acidosis. Investigators will know specific brain areas related to sng perception evoked by the peripheral muscle acidosis and, accordingly, a novel mechanism and potential treatment for sng would be developed in this proposed study.

DETAILED DESCRIPTION:
Sng is a prominent complaint in Taiwanese people with low back pain. "Sng" is created to represent this Taiwanese word. Based on investigators preliminary data, sng was one of the most common complaints in patients with chronic low back pain (CLBP) and also one of the most common indication for lumbar spine operations. Back sng is not adequately relieved by pain-killers or even by the lumbar spine operations. By using functional magnetic resonance imaging and questionnaires, the investigators preliminary study demonstrated that sng is different from pain in the level of brain perception and the level of subjective concept. It is very likely that sng has its own unique nerve pathway other than pain. The subjective feeling of sng is very similar to sour in taste, so it is likely that acidosis may be involved in the process of sng sensation, especially in the muscle. Delayed onset muscle soreness is a well-known example, and the soreness is dependent on the proton-sensing neurons. Indeed, substantial evidences showed that up to 80% muscle afferents are acid-sensitive but not nociceptors. Therefore, the investigators propose that sng is the perception in the brain when the tissue acidosis is sensed by the somatosensory system, and "sng-ception" is created to indicate the sensation of tissue acidosis. However, the causal connection between the peripheral sngception and the central brain perception of sng is not established. The objective of this proposal is to establish the causal connection between peripheral muscle acidosis and the central brain sng perception. The investigators central hypothesis is that acidosis-evoked sensation in the muscles will cause a central sng perception in the brain. This hypothesis is based on investigators previous studies that showed sng is different from pain in terms of subjective responses, brain activation areas and clinical impacts. To achieve this goal, two specific aims will be pursued 1. to determine if an acid solution will evokes sng response, and, 2. to detect the brain activation area of sng evoked by an acid solution in functional magnetic resonance imaging. Successful establishment of the casual connection between the peripheral muscle acidosis and the central brain sng perception will lead to a more comprehensive understanding of sng mechanism and the potential medication development.

ELIGIBILITY:
Inclusion Criteria:

1. The subject ages ranges from 20-45 years old.
2. The subject has no chronic pain symptoms or complaint in last 6 months.
3. The subject is subjectively able to discriminate sng and pain.
4. The subject has no history of major diseases that required treatment or currently being under treatment.
5. Gender: men and women half
6. The used hand of subject is the right hand.
7. The educational level of subject is more than 9 years (graduated from junior high school)
8. The subject didn't have physical and mental illness
9. The subject didn't take prescribed medicine.
10. The VAS questionnaire must be 0 point both of low back "pain" and low back "soreness" assessment.
11. The subject who can fill the informed consent after understanding the purpose and medical help of this trial.

Exclusion Criteria:

1. The subject has: Neuropathic pain due to causes other than that specified in the inclusion criteria (e.g., post-herpetic neuralgia; painful diabetic neuropathy; mononeuritis multiplex; central poststroke pain; failed back surgery in relation to the presenting episode of radiculopathy; spinal abscess, infection, hematoma, or malignancy; phantom limb pain; peripheral neuropathy due to alcoholism, malignancy, human immunodeficiency virus [HIV], syphilis; drug abuse; vitamin B12 deficiency; hypothyroidism; liver disease; toxic exposure). Pain that is associated with a substantial somatic pain component (e.g., non-neuropathic/musculoskeletal pain in lower limbs or other parts of the body apart from the back) or more than one cause or potential cause for pain symptoms.Any painful concurrent rheumatic disease such as, but not limited to, fibromyalgia, rheumatoid arthritis, or significant osteoarthritis.
2. The subject is unable to reliably delineate or assess his or her own pain by anatomical location/distribution (e.g., the subject cannot reliably tell the difference between his or her back pain and lower limb pain and cannot rate the intensity of each separately).
3. The subject has undergone lumbar spine surgery within the last 6 months or has received treatment with epidural injections, nerve blocks, or acupuncture for lower skin electrical resistance within 4 weeks before screening.
4. The subject had a malignancy according to his/her report.
5. The subject had allergic to lidocaine or monobasic sodium phosphate and dibasic sodium phosphate
6. The subject has had a positive test for HIV antibody or a history of HIV according to his/her report.
7. The subject has had a positive test for hepatitis B surface antigen or hepatitis C antibody according to his/her report.
8. The subject has a history of alcohol or narcotic substance abuse according to his/her report.
9. The subject is female and is pregnant or breastfeeding at the time of the screening visit or plans to become pregnant during the study period.
10. The subject cannot perform brain MRI scanning who had metal implants of head (such as fixed dentures, metal bone plate, vascular clamp, vascular embolization treatment coil, deep brain stimulator, artificial electronic ear, etc.), implants of head which affecting the image quality (such as the ventricle peritoneal catheter, etc.), implantation of permanent heart rate regulator, etc.
11. The subject has suffered from claustrophobia.
12. The subject has a history of spinal surgery.
13. The VAS questionnaire not be 0 point either low back "pain" or low back "soreness" assessment.
14. The subject has mental comorbidity (such as depression, panic disorder, etc)
15. The subject has suffered from brain disease and had brain surgery.
16. The subject has taken prescribed medicine which can affect specific function of brian (such as sleeping pills, tranquilizer, etc.).
17. The subject has mental retardation.
18. The educational level of subject is less than 9 years.
19. The subject who under 20 years old or older than 45 years old, who is unable to understand the purpose of this trial and fill the informed consent.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2019-07-11 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Brain functional magnetic resonance imaging | The whole procedures will be done within 50 minutes. Before the injection, the subject will receive anatomical MRI scan (10 minutes) and baseline fMRI scan (10 minutes) After that, the acid or pH 7.4 PBS will be given into the midpoint of the left tibial
  All images will be acquired on a 3 Tesla MRI system (MAGNETOM Prisma, Siemens, Erlangen, Germany) with a 20-channel head coil. To obtain an anatomical reference, high-resolution T1-weighted imaging was performed using a 3D magnetization-prepared rapid gradient echo (MPRAGE) sequence: repetition time (TR)/echo time (TE) = 2000 ms/3 ms, flip angle = 9°, field of view (FOV) = 256 × 192 × 208 mm3, acquisition matrix = 256 × 192 × 208, resulting in isotropic spatial resolution of 1 mm3. The task fMRI will be performed using an echo planar imaging (EPI) sequence with a twice-refocused balanced echo. The imaging parameters are: TR/TE = 2000/20 ms, slice thickness = 3.5 mm, 80 × 80 acquisition matrix, FOV = 200 × 200 mm, and in-plane spatial resolution = 3.0 mm x 3.0 mm.

SECONDARY OUTCOMES:
The visual analog scale (VAS) of "sng" in the legs | Through fMRI completion an average of 6 months
  The subject will be asked for sng VAS before infusion and immediately after infusion.
  Scale range 0 to 10 (1)0: No Sng (2)1-3: Mild Sng (3)4-6: Moderate Sng (4)7-9: Severe Sng (5)10: Worst Sng imaginable
Muscle pressure pain threshold | Through fMRI completion an average of 1 week
  Muscle pressure pain threshold on bilateral tibialis anterior muscles will be measured by algometer.

OTHER OUTCOMES:
36-Item Short Form Health Survey (RAND) | Up to 6 months before signing the informed consent form
  Investigator will evaluate the subject life quality and activity of daily life by 36-Item Short Form Health Survey (RAND) Consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
The visual analog scale (VAS) of "sng" in the back | Through fMRI completion an average of 6 months
  The subject will be asked for sng VAS before infusion and immediately after infusion.
  Scale range 0 to 10 (1)0: No Sng (2)1-3: Mild Sng (3)4-6: Moderate Sng (4)7-9: Severe Sng (5)10: Worst Sng imaginable
Oswestry disability index | Up to 6 months before signing the informed consent form
  Investigator will evaluate the subject activity of daily life by Oswestry disability index The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100) (1)0 -20: Minimal disability (2)21-40: Moderate Disability (3)41-60: Severe Disability (4)61-80: Crippling back pain (5)81-100: These patients are either bed-bound or have an exaggeration of their symptoms
The Hospital Anxiety and Depression Scale | Up to 6 months before signing the informed consent form
  Is a 14-item measure designed to assess anxiety and depression symptoms in subjects, with emphasis on reducing the impact of physical illness.
  Total score (Depression、Anxiety):
  (1)0-7 Normal (2)8-10 Borderline abnormal (borderline case) (3)11-21 Abnormal (case)
Edinburgh Handedness Inventory | Up to 6 months before signing the informed consent form
  Is a measurement scale used to assess the dominance of a person's right or left hand in everyday activities, sometimes referred to as laterality. The inventory can be used by an observer assessing the person.
  Handedness score is calculated using this formula: 100*((Right - Left) / (Right + Left)).
  1. Pure left hander: total score=-100
  2. Mixed left hander:-100< total score <0
  3. Neutral: total score=0
  4. Mixed right hander:0< total score <100
  5. Pure left hander:total score=100

CONTACTS AND LOCATIONS:
Overall Officials: Jiann-Her Lin, MD/PhD, Principal Investigator — Taipei Medical University Hospital
Locations (1):
- Taipei Medical University Hospital, Taipei, No.252, Wusing St., Sinyi Dist., Taiwan

REFERENCES:
- [Background] Issberner U, Reeh PW, Steen KH. Pain due to tissue acidosis: a mechanism for inflammatory and ischemic myalgia? Neurosci Lett. 1996 Apr 26;208(3):191-4. doi: 10.1016/0304-3940(96)12576-3. PMID 8733302
- [Background] Law LAF, Sluka KA, McMullen T, Lee J, Arendt-Nielsen L, Graven-Nielsen T. Acidic buffer induced muscle pain evokes referred pain and mechanical hyperalgesia in humans. Pain. 2008 Nov 30;140(2):254-264. doi: 10.1016/j.pain.2008.08.014. Epub 2008 Oct 2. PMID 18835099
- [Background] Lin JH, Hung CH, Han DS, Chen ST, Lee CH, Sun WZ, Chen CC. Sensing acidosis: nociception or sngception? J Biomed Sci. 2018 Nov 29;25(1):85. doi: 10.1186/s12929-018-0486-5. PMID 30486810
- [Background] Fujii Y, Ozaki N, Taguchi T, Mizumura K, Furukawa K, Sugiura Y. TRP channels and ASICs mediate mechanical hyperalgesia in models of inflammatory muscle pain and delayed onset muscle soreness. Pain. 2008 Nov 30;140(2):292-304. doi: 10.1016/j.pain.2008.08.013. Epub 2008 Oct 1. PMID 18834667
- [Background] Chen CC, Wong CW. Neurosensory mechanotransduction through acid-sensing ion channels. J Cell Mol Med. 2013 Mar;17(3):337-49. doi: 10.1111/jcmm.12025. Epub 2013 Mar 14. PMID 23490035
- [Background] Chen WN, Lee CH, Lin SH, Wong CW, Sun WH, Wood JN, Chen CC. Roles of ASIC3, TRPV1, and NaV1.8 in the transition from acute to chronic pain in a mouse model of fibromyalgia. Mol Pain. 2014 Jun 23;10:40. doi: 10.1186/1744-8069-10-40. PMID 24957987